CLINICAL TRIAL: NCT00822913
Title: The Use of Toxin Botulinum A Toxin in Patients With Parkinson's Disease and Multiple System Disease, Affected by Refractory Detrusor Overactivity.
Brief Title: Botulinum A Toxin in Patients With Parkinson's Disease
Acronym: Botox-PD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Of Perugia (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Giannantoni Antonella, University of Perugia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-B-PD
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2009-01-15 (Estimated); Status verified 2009-01

CONDITIONS: Parkinson's Disease; Multiple System Atrophy; Detrusor Overactivity
Keywords: Botulinum A toxin; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Urinary Bladder, Overactive | interventions — Idoxuridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Botulinum A toxin (Experimental): Botulinum A toxin intravesical injection
  Interventions: Drug: Intravesical injection of Botulinum A toxin

INTERVENTIONS:
Drug: Intravesical injection of Botulinum A toxin — One treatment, 200 U vials diluted in 20 ml normal saline
  Other Names: Allergan

SUMMARY:
The researchers investigated the effectiveness and safety of BoNT/A injected into the detrusor muscle in patients with PD and MSA all of whom had detrusor muscle overactivity unresponsive to conventional medical therapy.

DETAILED DESCRIPTION:
Patients included will have overactive bladder symptoms refractory to medical therapy. Other causes of overactive bladder symptoms including urogenital prolapse and recurrent urinary tract infections were excluded. None of the patients will be under anticoagulant therapy or drugs interfering with neuromuscular transmission. The study was approved by the local ethical committee and patients gave their informed consent. Patients will be informed about the possible need for intermittent catheterization after BoNT/A treatment.

As outcome measures we assessed clinical and urodynamic variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients with overactive bladder symptoms refractory to medical therapy.

Exclusion Criteria:

* Other causes of overactive bladder symptoms including urogenital prolapse and recurrent urinary tract infections were excluded.
* Concomitant anticoagulant therapy or drugs interfering with neuromuscular transmission.
* Neuromuscular disease like Lambert-Eaton syndrome.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
As primary outcome measures, patients attended for clinical evaluation (daily voiding diary an QoL questionnaire). | One, three and five months after intravesical treatment

SECONDARY OUTCOMES:
Urodynamic assessment, and samples were obtained for urinalysis and culture. | One, three and five months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Giannantoni, M.D., Principal Investigator — University Of Perugia